CLINICAL TRIAL: NCT06710743
Title: Determination of the Glycemic Index Values of 10 Cereal-based Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2402
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Low Glycemic Index (GI) Food; Pre Diabetes; Diabetes
Keywords: Low GI food; glycemic index; cereal; carbohydrate; glucose
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Reference food (Active Comparator): Glucodin powder solution
  Interventions: Other: Glucose solution Day 1, Day 8, and Day 15
- Food 1 (Experimental): Quaker Whole Oats
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 2 (Experimental): Quaker Quick Cooking White Oats
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 3 (Experimental): Saffola Oats
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 4 (Experimental): Quaker Oats
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 5 (Experimental): Quaker Oats Multigrain
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 6 (Experimental): Ragi Flakes
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 7 (Experimental): Bajra Flakes
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 8 (Experimental): Jowar Flakes
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 9 (Experimental): Maltabella
  Interventions: Other: Food (cereal). Ten different cereals served once each
- Food 10 (Experimental): FutureLife Smart + White Oats
  Interventions: Other: Food (cereal). Ten different cereals served once each

INTERVENTIONS:
Other: Glucose solution Day 1, Day 8, and Day 15 — Glucodin powder diluted with water
  Arms: Reference food
Other: Food (cereal). Ten different cereals served once each — Variety of cooked or flake cereal
  Arms: Food 1; Food 10; Food 2; Food 3; Food 4; Food 5; Food 6; Food 7; Food 8; Food 9

SUMMARY:
To determine the Glycemic index values for 10 cereal-based products

DETAILED DESCRIPTION:
To determine the Glycemic index values for 10 cereal-based products per international standard (ISO26642:2010) for glycemic index determination.

ELIGIBILITY:
Inclusion Criteria:

* 10 healthy participants, male and female (non-pregnant, non-lactating) of mixed ethnicity, aged between 18 - 65 y
* BMI: 18 - 25.0 kg/m2 (bounds included)
* Non smokers
* Normal glucose tolerance (assessed by 50 gram oral glucose tolerance test performed within the last 30 days: fasting <6 mM, 2 hr glucose <7.8 mM)
* Stable weight and dietary habits. Normal eating patterns and no history of eating disorders or recent dieting
* Normal sleep patterns (ie. at least 6 hours of sleep per night)
* The participants are required to avoid alcohol and unusual levels of food intake and physical activity for the 24 hours before each test session.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history. Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Food allergy or intolerance to the study ingredients (eg. gluten, etc.)
* Regularly taking prescription medication other than standard contraceptive medication
* Taking any medications known to affect glucose tolerance (eg. acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis)
* Suffering from any illness or disease
* Following a restricted diet
* Smokers
* Eating disorders
* Abnormal glucose tolerance or known history of diabetes mellitus.
* Individuals currently participating in other acute metabolic studies
* Failure to meet any one of the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Glycemic index (GI) values | Two hour test session per visit. Visits must be at least two days apart. Including Screening, the study duration is approximately four to eleven weeks depending on whether participants are available to be tested one, two or three times per week.
  Comparison of Glycemic index (GI) values of 10 different cereal-based products and the reference food (glucose solution assigned GI=100 by definition)

CONTACTS AND LOCATIONS:
Overall Officials: Richa Bharti, MS, Principal Investigator — PepsiCo R&D Life Sciences
Locations (1):
- Sydney University's Glycemic Index Research Service (SUGiRS), Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No